CLINICAL TRIAL: NCT07104162
Title: A Phase 1, Open-label, Single-dose Study to Determine the Safety and Pharmacokinetics of Intravenous Cefiderocol/Xeruborbactam (S-649228) in Participants With Renal Impairment
Brief Title: A Study to Investigate Safety and Pharmacokinetics of Intravenous Cefiderocol/Xeruborbactam in Participants With Renal Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qpex Biopharma, Inc. (Industry)
Collaborators: Shionogi Inc. (Industry); Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Qpex-401
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Bacterial Infections
Keywords: beta-lactamase inhibitor
MeSH Terms: conditions — Bacterial Infections | interventions — Cefiderocol; QPX7728

STUDY DESIGN:
Intervention Model Description: Open-label, single-dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label, Single Dose of IV Cefiderocol/Xeruborbactam (Experimental): Approximately 40 participants will be enrolled in total. Eight participants will be enrolled in each group (G) based on renal impairment (RI) determined by estimated glomerular function rate (eGFR) or need for intermittent hemodialysis (IHD) at screening:
  * G1: Mild RI (eGFR 60 < 90 mL/min calculated using the 2021 Chronic Kidney Disease Epidemiology Collaboration equation [CKP-EPI]) adjusted for the participant's body surface [BSA])
  * G2: Moderate RI (eGFR 30 to < 60 mL/min calculated using the 2021 CKD-EPI equation adjusted for the participant's BSA)
  * G3: Severe RI (eGFR < 30 mL/min calculated using the 2021 CKD-EPI equation) not receiving IHD therapy
  * G4: Healthy participants with normal renal function matched to participants in Groups 1 and 2 (Group 3 may be included) based on age, gender and body mass index (BMI)
  * G5: Participants with end stage renal disease (ESRD) receiving IHD
  All participants will receive a single dose of cefiderocol/xeruborbactam on Day 1.
  Interventions: Drug: Cefiderocol/Xeruborbactam

INTERVENTIONS:
Drug: Cefiderocol/Xeruborbactam — A fixed dose combination of intravenous cefiderocol and intravenous xeruborbactam
  Other Names: Cefiderocol/QPX7728; S-649228

SUMMARY:
A Phase 1, Open-label, Single-dose Study to Determine the Safety and Pharmacokinetics of Intravenous Cefiderocol/Xeruborbactam (S-649228) in Participants with Renal Impairment

DETAILED DESCRIPTION:
Qpex Biopharma, Inc., a wholly owned subsidiary of Shionogi Inc., is developing a fixed combination antibiotic of cefiderocol, a cephalosporin antibiotic approved in the US for the treatment of complicated urinary tract infections (cUTIs) including pyelonephritis, and hospital-acquired bacterial pneumonia (HABP) and ventilator-associated bacterial pneumonia (VABP), plus an investigational broad-spectrum beta-lactamase inhibitor (BLI), xeruborbactam (QPX7728) to address the need for new antibiotics for the pathogens deemed as urgent or critical threats.

The aim of this study is to compare single-dose intravenous (IV) pharmacokinetics (PK) and safety of the combination of cefiderocol/xeruborbactam (S-649228) in participants with various degrees of stable renal impairment, including those with end-stage renal disease (ESRD), to control participants with normal renal function.

The results from this study will enable the development of appropriate dosing recommendations in patients with impaired renal function.

Objectives:

The objectives of the study are:

1. To assess the impact of mild, moderate, and severe renal impairment, and intermittent hemodialysis (IHD) on the PK of IV cefiderocol and IV xeruborbactam given to participants with stable renal impairment, normal renal function, and ESRD receiving IHD therapy.
2. To evaluate the safety and tolerability of IV cefiderocol and IV xeruborbactam given to participants with stable renal impairment, normal renal function, and ESRD receiving IHD therapy.

ELIGIBILITY:
Inclusion Criteria:

An individual will be eligible to be included in the study only if all of the following criteria apply:

All participants

* Able to understand the study conduct and tasks required of the participants, sign the informed consent form and willing to cooperate with all tests and examinations required by the protocol.
* Aged 18 to 80 years, inclusive, at the time of consent.
* If male, agrees to be sexually abstinent or agrees to use 2 approved methods of contraception (refer to Inclusion Criterion 4) when engaging in heterosexual activity from Day -1 through 90 days following the last administration of the study intervention, and to not donate sperm during this same period of time. If the sexual partner is surgically sterile, contraception is not necessary.
* If female of childbearing potential, must either be sexually abstinent for 14 days prior to Day -1 and remain so through 30 days following dosing of the study intervention or have been using (or agree to use) 2 acceptable methods of birth control when engaging in heterosexual activity
* If female of childbearing potential, must agree not to donate eggs (ova, oocytes) for the purpose of reproduction from Day -1 through 30 days following the last administration of the study intervention.
* If female of non-childbearing potential, must either be postmenopausal (defined as 12 months spontaneous amenorrhea) with serum follicle stimulating hormone (FSH) level in the laboratory-defined postmenopausal range or have undergone sterilization procedures at least 6 months prior to Day -1; documentation of sterilization procedure must be obtained
* Has a BMI ≥ 18.5 kg/m2 and ≤ 45 kg/m2, inclusive.
* Has negative test results for hepatitis B surface antigen (HBsAg), anti-Hepatitis C virus (HCV) antibody, anti-human immunodeficiency virus (HIV) antibody, and SARS-CoV-2.

Participants with normal renal function:

* Has an eGFR ≥ 90 mL/min calculated using the 2021 CKD-EPI equation adjusted for the participant's BSA at screening
* Meets matching criteria for age, BMI, and gender of pooled renally impaired participants as defined in the protocol.

Participants with renal impairment

* Stable mild to severe renal impairment, as assessed by eGFR calculated using the 2021 CKD-EPI equation adjusted for the participant's BSA at screening
* Is on a stable medication regimen

Participants with ESRD on hemodialysis

* Receiving stable IHD at least 3 times a week for at least 3 months, using an arteriovenous fistula, graft, or catheter
* Is on a stable medication regimen

Exclusion Criteria:

An individual must not meet any of the following exclusion criteria to be eligible to participate in the study:

* Has unstable or new medical condition(s)
* Has had surgery under general anesthesia within the past 3 months prior to Day -1, determined by the investigator to be clinically relevant.
* Documented hypersensitivity reaction or anaphylaxis to any medication.
* History of seizures, convulsions
* Current evidence or history of malignancy
* If female, is pregnant, lactating, or has a positive pregnancy test at screening or Day -1.
* Received any investigational drug within 30 days or 5 half-lives, whichever is longer, of Day -1 for the current clinical study.
* Blood donation or significant blood loss (ie, > 500 mL) within 56 days prior to Day -1.
* Plasma or platelet donation within 14 days prior to Day -1.
* Any acute illness requiring antibiotic drug therapy within 30 days prior to Day -1 or a febrile illness within 7 days prior to Day -1.
* Vigorous exercise from 72 hours prior to Day -1 through the final FU/EOS Visit.
* Positive drug test at the Screening Visit or Day -1
* Positive alcohol test at screening or Day -1 and/or recent history (ie, within 6 months prior to Day -1) of excessive alcohol intake.
* Concurrent use of medications known to affect the elimination of serum creatinine and competitors of renal tubular secretion
* Employees of the investigative site involved in this study.
* Unable or unwilling to adhere to the study-specified procedures and restrictions.
* QTcF interval > 500 msec, previous history or family history of prolonged QT syndrome at screening or Day -1.
* Use of products containing alcohol, caffeine, xanthine, or ephedrine within 24 hours prior to Day -1; use of alcohol 48 hours prior to Day -1; use of proton pump inhibitors (eg, omeprazole and pantoprazole) 7 days prior to Day -1, including both over-the-counter (OTC) and prescription drugs in these categories; or consumption of grapefruit/grapefruit juice, Seville oranges, pomelo, exotic citrus fruits or grapefruit hybrids or juices containing such products within 7 days prior to Day -1.
* Has any clinically significant abnormalities in laboratory values at screening or Day -1, defined in the study protocol.

Participants with normal renal function:

• Abnormal and clinically significant findings on physical examination, medical history, serum chemistry, hematology, or urinalysis per Investigator discretion.

Participants with renal impairment, including those on IHD:

* Abnormal and clinically significant findings on physical examination, medical history, serum chemistry, hematology, or urinalysis per Investigator discretion. Participants in the renal impairment group will have consideration for the degree of renal impairment and presence of comorbidities.
* Has renal disease secondary to hepatic disease (hepatorenal syndrome)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) by participant and by group | 11-22 days (+/- 2)
  Number of participants with treatment-emergent adverse events by severity and relationship to treatment
Number of participants with changes from baseline in safety parameters | 11-22 days (+/- 2)
  Number of participants with changes in safety parameters before and after dosing by subject and group
Maximum plasma concentration measurements by subject and by group (Cmax) | 11-22 days (+/- 2)
  Comparison will be performed between the groups for maximum plasma concentration (Cmax).
Time to maximum plasma concentration (Tmax) | 11-22 days (+/- 2)
  Comparison will be performed between the groups for time to maximum plasma concentration (Tmax)
Area under the plasma concentration versus time curve (AUC) | 11-22 days (+/- 2)
  Comparison will be performed between the groups for area under the plasma concentration versus time curve (AUC)
Cumulative amount of drug excreted as unchanged in the urine (Aeu) | 11-22 days (+/- 2)
  This parameter will not be estimated in Group 5
Cumulative amount of drug excreted as unchanged in the dialysate (Aed) | 11-22 days (+/- 2)
  This parameter will be estimated only in Group 5. Urine pharmacokinetic (PK) parameters will be calculated from urinary excretion and dialysate data.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Richard Preston, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No